CLINICAL TRIAL: NCT04531111
Title: Glycemic Control Among Children and Adolescents With Type 1 Diabetes During COVID-19 Pandemic in Egypt: A Pilot Study
Brief Title: Glycemic Control Among Children and Adolescents With Type 1 Diabetes During COVID-19 Pandemic in Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasmine Ibrahim Elhenawy, Assistant Professor of Pediatrics, Ain Shams University
Other Study IDs: FMASU P66/2020
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Type 1 Diabetes; Covid19
Keywords: Type 1 Diabetes; Glycemic control; COVID-19
MeSH Terms: conditions — Diabetes Mellitus, Type 1; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the current unusual situation with COVID-19 pandemic and the lockdown applied in most of the countries, school students were kept at home and offered e-learning modules and all activities were suspended.

Lockdown entails significant modifications of life style, involving changes in physical activities, dietary habits and nutrition, which are likely to impact glycemic control.

So the aim of the current study is to evaluate the impact of COVID-19 pandemic on glycemic control among children and adolescents with type 1 diabetes.

DETAILED DESCRIPTION:
All aspects of life were significantly impacted by the COVID-19 pandemic. The pandemic created heavy burdens on all countries affecting all foundations of the country. Global measures aimed to limit spread of COVID- 19 infection and a series of restriction were announced by serial countries including the suspension of schools, organized sports activities and gatherings. On March, 2020 Egypt started to take a series of lockdown regulation to control the spread of infection.

The restriction and lockdown will impact the whole population especially populations with chronic disease. It is known that the lockdown will render access to outpatient clinics and services,beside the possible limitation of access to care, the restrictions may affect glycemic control patients with diabetes.

The negative impact of limiting physical exercise, behavioral changes, dietary changes and fear of shortage of medical supplies could have an influence on diabetes control.

Study procedure:

All included patients / caregivers will complete an online questionnaire. For patients with limited internet access, the questionnaire will be carried out through phone calls according to patients' convenience.

Perceived stress scale-10 (Arabic Validated version) will be used to measure patients'/ caregivers' level of stress in response to the extraordinary status of the pandemic and its consequences. The scale is a 10 questions scale that will be circulated among the patients as an Arabic validated electronic form .

Medical reports and files of included patients will be reviewed and last visit before the lock down will be thoroughly evaluated to identify:

* Patients' body weight, body mass index.
* Insulin regimen with special emphasis on total daily dose and percentage of basal insulin.
* Glycemic control of patients by evaluating the last HbA1C After completing the questionnaire, patients' insulin dosage and glycemic control during the quarantine period will be re-evaluated.

Evaluation of glycemic control at the end of the study:

* For patients on self- monitoring of blood glucose, a rapid Hba1c test will be done according to patients' convenience, patterns and frequency of hypoglycemia and hyperglycemia will be evaluated.
* For those on continous glucose monitoring ( if available), the data will be extracted from the ambulatory glucose profile(AGP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes and willing to participate in the study.
* Age: less than 18 years old

Exclusion Criteria:

* Newly diagnosed patients with type 1 diabetes and those in honeymoon period.
* Children with other forms of diabetes, including: type 2, monogenic forms and secondary diabetes.
* Patients with any other chronic disease.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Data will be collected from patients who are conveniently available and willing to participate in the study in the period from July to August 2020, will be used. A questionnaire will be circulated among patients and/or their caregivers and can be filled online or through telephone calls.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Impact of COVID-19 pandemic and lockdown on glycemic control among a sample of Egyptian children and adolescents with type 1 diabetes | 12 weeks
  Change in HbA1c from baseline to 3 month after the lockdown

SECONDARY OUTCOMES:
Impact of COVID-19 pandemic and lockdown on insulin dosage among a sample of Egyptian children and adolescents with type 1 diabetes | 12 weeks
  Change in total insulin dosage from baseline to 3 month after the lockdown

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine Elhenawy, Principal Investigator — Ain Shams University
Locations (1):
- Pediatrics and Adolescents Diabetes Unit (PADU), Pediatrics Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided